CLINICAL TRIAL: NCT02573298
Title: Cryotherapy and Doppler in Inflammatory Rheumatic Diseases
Acronym: CDRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); Groupement Interrégional de Recherche Clinique et d'Innovation (Other); Etablissement Français du Sang (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P/2012/148
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis; Crystal-induced Arthritides; Spondyloarthritis
Keywords: cryotherapy; power Doppler score; synovial fluid cytokines; pain VAS
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis | interventions — Dental Pulp Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ice (Active Comparator): patients randomized to receive local ice on inflamed joint
  Interventions: Device: ice
- Cold gas (Active Comparator): patients randomized to receive cold gas on inflamed joint
  Interventions: Device: cold gas

INTERVENTIONS:
Device: ice — local ice application for 30 minutes
  Other Names: ice pack
  Arms: Ice
Device: cold gas — local cold gas application for 2 minutes
  Other Names: Cryo+ (pulsed hyperbaric CO2)
  Arms: Cold gas

SUMMARY:
The primary aim of the study is to evaluate the effects of two local cryotherapy (ice or cold gas) applications on arthritic knees.

Evaluation criteria (before/after treatment):

* synovial power-Doppler semi-quantitative score
* pain VAS (mm)
* cytokine levels in synovial fluid
* leukocyte count in synovial fluid

DETAILED DESCRIPTION:
After informed consent, patients suffering from inflammatory rheumatic diseases (rheumatoid arthritis, spondyloarthritis, crystal-induced arthritides) with non-septic arthritides were randomized to receive either local ice (30 minutes twice a day) or cold gas (2 minutes twice a day - pulsed hyperbaric CO2). Local cryotherapy was applied at 9 AM and 17 PM.

Skin temperature was monitored Knee power Doppler ultrasonography was performed before cryotherapy (9 AM), just after, 2 min after, 2 hours after, before and after the second cold application (8 hours after the first cold application), then the day after at 9 A.M (24 hours after the first cold application).

Synovial fluid was also analysed after join arthrocentesis (just before the first cold application, then 24 hours later, after the last ultrasonographic examination. A corticosteroid injection was performed after the second arthrocentesis when necessary.

Power Doppler semi-quantitative scores (0-3) were then blindly assessed by a second trained ultrasonographist at the different times of the study.

Pain VAS evolution was also monitored throughout the study. Clinical characteristics of patients were collected at baseline. 20 patients suffering from ankle/wrist arthritides were also included in order to evaluate power Doppler score evolution under cold gas or ice-cryotherapy.

15 patients suffering from knee arthritides were treated by local cold gas. 31 patients suffering from knee arthritides were treated by ice. When both knees were arthritic, contralateral synovial fluid and power Doppler score were used as non-treated controls.

ELIGIBILITY:
Inclusion Criteria:

* non-septic joint arthritis with power Doppler activity( score>=1/3)

Exclusion Criteria:

* neurologic diseases impairing skin sensitivity
* cold allergia
* Raynaud phenomenon
* non-controlled diabetes mellitus, heart failure, heart pace abnormalities
* skin lesion on the application area
* cognitive impairments
* active vasculitis
* paroxystic haemoglobinuria
* cryoglobulin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02; Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Power Doppler score change (Naredo's 0-3 semi-quantitative scale) | Baseline, 2 minutes, 2 hours, 8 hours, 24 hours
  Semi-quantitative power Doppler score was assessed at baseline, just after, 2 min after, 2 hours after, 8 hours after (just before the second cold application then just after), 24 hours after the first cold application.
IL-6 levels in knee synovial fluid change (Multiplex, cytometry) | Baseline, 24 hours
  synovial fluid was analysed at baseline, then 24 hours later (after the last ultrasonographic examination)

SECONDARY OUTCOMES:
pain VAS change (numeric scale) | Baseline, 2 minutes, 2 hours, 8 hours, 24 hours
  pain VAS (mm) was recorded at each ultrasonographic examination
synovial fluid leukocyte count change (per mm3) | Baseline, 24 hours
IL-1beta, TNF-alpha, IL-17, VEGF level changes in the synovial fluid (Multiplex, cytometry) | Baseline, 24 hours
skin temperature change (°C, skin temperature probe in the application area) | Baseline, 2 minutes, 2 hours, 8 hours, 24 hours
  Skin temperature will be measured during each ultrasonographic examination

CONTACTS AND LOCATIONS:
Overall Officials: Xavier GUILLOT, MD, Principal Investigator — Centre Hospitalier Universitaire de Besançon
Locations (1):
- Centre hospitalier universitaire de Besançon, Besançon, Franche-Comté, France

REFERENCES:
- [Result] Guillot X, Tordi N, Mourot L, Demougeot C, Dugue B, Prati C, Wendling D. Cryotherapy in inflammatory rheumatic diseases: a systematic review. Expert Rev Clin Immunol. 2014 Feb;10(2):281-94. doi: 10.1586/1744666X.2014.870036. Epub 2013 Dec 18. PMID 24345205
- [Derived] Guillot X, Tordi N, Prati C, Verhoeven F, Pazart L, Wendling D. Cryotherapy decreases synovial Doppler activity and pain in knee arthritis: A randomized-controlled trial. Joint Bone Spine. 2017 Jul;84(4):477-483. doi: 10.1016/j.jbspin.2016.09.004. Epub 2016 Nov 4. PMID 27825572